CLINICAL TRIAL: NCT00218842
Title: Physical and Daily Activity for Residents in a Nursing Home Setting. -A Nordic Multi-Centre Study
Brief Title: The Effect on Function of Increasing Activity for Nursing Home Residents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Helse Midt-Norge (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 203-04
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2014-03-07 (Estimated); Status verified 2014-03

CONDITIONS: Frailty; Nursing Home Residents
Keywords: exercise; functioning; frail elderly
MeSH Terms: conditions — Frailty; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- exercise group (Experimental): individualized exercise
  Interventions: Behavioral: Individualized exercise
- control group (No Intervention): care as usal

INTERVENTIONS:
Behavioral: Individualized exercise — individualized exercise, physical activity and training in daily life situations given by trained physical therapists and occupational therapists
  Arms: exercise group

SUMMARY:
As designs of existing outcome studies are disparate and do not always relate well to a Swedish context, the need for further studies is obvious. Also, an empirical theory drawn from the best practice supporting autonomy and wellbeing for clients in a nursing home setting has not yet been fully depicted. The study described below intends to fill a gap in knowledge related to the effect of enhanced activities of daily living (ADL)-training, physical, and daily activities and staff education in a nursing home setting, based on a theory- and evidence-based intervention programme in a Swedish as well as a Nordic health care context. The aims of the study are to describe the impact of an individually tailored intervention program, in a nursing home setting, on:

* Physical capacity
* Degree of dependence in ADL
* Long-term participation in physical and/or daily activities
* Self-rated wellbeing

DETAILED DESCRIPTION:
The Trondheim study has additional aims to assess the impact of intervention on:

* Urinary incontinence
* Falls

ELIGIBILITY:
Inclusion Criteria:

* > 65 years of age
* Expected stay in the nursing home > 3 months
* Able to take instruction

Exclusion Criteria:

* Persons in a terminal phase

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 125 (Actual)
Dates: Start 2005-10; Primary Completion 2009-10 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Physical function | baseline, three and six months

SECONDARY OUTCOMES:
Falls | during six months

CONTACTS AND LOCATIONS:
Overall Officials: Jorunn L Helbostad, PhD, Study Chair — St. Olavs University Hospital and Norwegian University of Science and Technology
Locations (1):
- Section of Geriatric Medicine, St. Olavs University Hospital, Trondheim, Trondheim, Norway

REFERENCES:
- [Background] Frandin K, Borell L, Gronstedt H, Bergland A, Helbostad JL, Puggaard L, Andresen M, Granbo R, Hellstrom K. A Nordic multi-center study on physical and daily activities for residents in nursing home settings: design of a randomized, controlled trial. Aging Clin Exp Res. 2009 Aug-Oct;21(4-5):314-22. doi: 10.1007/BF03324921. PMID 19959920
- [Background] Gronstedt H, Hellstrom K, Bergland A, Helbostad JL, Puggaard L, Andresen M, Granbo R, Frandin K. Functional level, physical activity and wellbeing in nursing home residents in three Nordic countries. Aging Clin Exp Res. 2011 Oct-Dec;23(5-6):413-20. doi: 10.1007/BF03337766. Epub 2011 Feb 10. PMID 21311211
- [Result] Gronstedt H, Frandin K, Bergland A, Helbostad JL, Granbo R, Puggaard L, Andresen M, Hellstrom K. Effects of individually tailored physical and daily activities in nursing home residents on activities of daily living, physical performance and physical activity level: a randomized controlled trial. Gerontology. 2013;59(3):220-9. doi: 10.1159/000345416. Epub 2012 Dec 20. PMID 23258191